CLINICAL TRIAL: NCT07343232
Title: Safety and Efficacy of Normobaric Facemask Oxygen for Hypocapnia in Aneurysmal Subarachnoid Hemorrhage(FOCAL): A Prospective, Multicenter, Proof-of-concept Pilot Study
Brief Title: Correcting Hypocapnia in Aneurysmal Subarachnoid Hemorrhage.
Status: Not yet recruiting | Type: Observational
Sponsor: The Chinese University of Hong Kong, Shenzhen (Other)
Responsible Party: Principal Investigator, Renzhi Wang, director of department, The Chinese University of Hong Kong, Shenzhen
Other Study IDs: CUHKShenzhen
Record Dates: First submitted 2025-12-17; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage (aSAH)
Keywords: Aneurysmal Subarachnoid Hemorrhage (aSAH); Hypocapnia
MeSH Terms: conditions — Subarachnoid Hemorrhage; Hypocapnia | interventions — Control Groups

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Normobaric Facemask Oxygen: Patients who received oxygen via a rebreathing facemask (ensuring no one-way valve is present), with a fractional inspired oxygen (FiO2) of 25-40% and an oxygen flow rate of ≤ 5 L/min.
  Interventions: Behavioral: Normobaric Facemask Oxygen
- Control group: Patients who received oxygen via nasal cannula or did not receive oxygen therapy.
  Interventions: Behavioral: control group

INTERVENTIONS:
Behavioral: Normobaric Facemask Oxygen — Oxygen is to be delivered via a rebreathing facemask (ensuring no one-way valve is present), with a fractional inspired oxygen (FiO2) of 25-41% and an oxygen flow rate of ≤ 5 L/min.
  The goals are to maintain patient SpO2 > 95%, PaCO2 between 35-42 mmHg, and, where feasible (particularly in centers with the capability for monitoring), an intracranial pressure (ICP) of < 15 mmHg.
  Groups: Normobaric Facemask Oxygen
Behavioral: control group — Using nasal cannula for oxygen inhalation or not using oxygen inhalation at all. Monitor and record the patient's SpO2, systolic blood pressure, diastolic blood pressure, PaCO2, and also monitor the intracranial pressure (ICP) at a center with monitoring capabilities.
  Groups: Control group

SUMMARY:
Based on the clinical observation that over half of the patients in the management of aneurysmal subarachnoid hemorrhage(aSAH) present with spontaneous hyperventilation, which is significantly associated with delayed cerebral ischemia and poor neurological outcomes, this prospective pilot study is designed to investigate the safety and efficacy of normobaric facemask oxygen for hypocapnia in aSAH.

DETAILED DESCRIPTION:
Spontaneous hyperventilation (SH) is highly prevalent following aneurysmal subarachnoid hemorrhage (aSAH) and is significantly associated with poor neurological outcomes.The core pathophysiological mechanism involves hypocapnia induced by hyperventilation, which triggers cerebral vasoconstriction and consequently leads to a decrease in cerebral blood flow (CBF).Although this response may transiently reduce intracranial pressure, persistent cerebral vasoconstriction markedly increases the risk of delayed cerebral ischemia (DCI) and secondary brain injury. Therefore, maintaining the arterial partial pressure of carbon dioxide (PaCO2) within the physiological range of mmHg is recommended to minimize the detrimental effects of hypocapnia.

Currently, there is a lack of standardized management strategies for hypocapnia resulting from SH after aSAH. Based on physiological principles, low-flow (<5 L/min) oxygen delivery via a facemask may effectively correct hypocapnia by promoting the rebreathing of carbon dioxide within the dead space of the facemask.10 A randomized controlled trial investigating psychogenic hyperventilation syndrome provides preliminary evidence for this approach, demonstrating that low-flow (3 L/min) facemask oxygen therapy can relieve symptoms more rapidly and improve patient comfort compared to traditional breathing training.11

However, high-level evidence regarding the safety, efficacy, and impact on neurological outcomes of using low-flow facemask oxygen therapy (functioning as a rebreathing mask) as a targeted intervention for correcting hypocapnia in aSAH patients remains scarce. Consequently, this proof-of-concept prospective study aims to systematically evaluate the operational safety and clinical effectiveness of rebreathing facemask oxygen therapy for correcting hypocapnia in patients with aSAH.

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years.
2. Confirmed diagnosis of aneurysmal subarachnoid hemorrhage (aSAH), with the presence of an aneurysm verified by computed tomography (CT), CT angiography (CTA), or digital subtraction angiography (DSA).
3. Hunt-Hess grade II-IV.
4. Presence of hypocapnia on arterial blood gas analysis, defined as PaCO2 < 35 mmH;
5. PaO2 > 90 mmHg.

Exclusion Criteria:

1. Presence of brain herniation or refractory intracranial hypertension, defined as a baseline intracranial pressure (ICP) > 25 mmHg that responds poorly to conventional ICP-lowering therapy;
2. Primary respiratory diseases (e.g., chronic obstructive pulmonary disease, severe asthma) known to cause chronically elevated baseline PaCO2;
3. Severe acid-base disturbances other than respiratory alkalosis.
4. Severe cardiac insufficiency, severe hepatic or renal dysfunction, malignant tumors, or other severe comorbidities that significantly impact prognosis;
5. Before the onset of the disease, the mRS score was greater than 2, and there were other factors causing disability.
6. Life expectancy < 3 months;
7. Any other condition deemed by the investigator to pose a high risk warranting exclusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Aneurysmal Subarachnoid Hemorrhage Patients with Hypocapnia.
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
modified Rankin Scale (mRS) >3 | 90-day follow-up visit
  The poor neurological outcome was considered to be mRs >3, indicating severe disability or death. The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. (Score Description: 0---No symptoms at all. 1---No significant disability despite symptoms; able to carry out all usual duties and activities. 2---Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance. 3---Moderate disability; requiring some help, but able to walk without assistance. 4--- Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance. 5---Severe disability; bedridden, incontinent and requiring constant nursing care and attention. 6---Dead.
Incidence of delayed cerebral injury (DCI) | 30 days after onset
  The presence of new focal neurological signs or a documented decrease in the level of consciousness persisting for at least 1 hour (or a drop of at least 1 point in the total Glasgow Coma Scale score), deemed to be of ischemic origin, after ruling out other causes (such as hydrocephalus, toxic-metabolic disturbances, or seizures); or identification of a new cerebral infarction on CT or MRI imaging.

SECONDARY OUTCOMES:
Montreal Cognitive Assessment (MoCA) | 90-day follow-up visit
  Cognitive function was evaluated using the Montreal Cognitive Assessment (MoCA), a standardized screening tool with scores ranging from 0 to 30, where higher scores indicate better cognitive performance and lower scores reflect greater cognitive impairment. Measure mean score or median compared between groups. And the rate of MoCA score of 20 or less between groups.
Cerebral Vasospasm | Participants will be followed for the duration of the hospital stay, an expected average of 2 weeks
  Incidence of moderate and severe radiographic cerebral vasospasm (catheter angiogram, CTA, MRA) or incidence OR moderate and severe vasospasm by transcranial doppler (TCD) criteria.
Glasgow Coma Score(GCS) | Enrollment, 30 days after onset, and 90-day follow-up visit
  The Glasgow Outcome Scale was used as secondary outcomes. The level of consciousness was assessed using the Glasgow Coma Scale (GCS), a standardized scale ranging from 3 to 15, where higher scores indicate a better neurological status (i.e., a higher level of consciousness), and lower scores reflect more severe impairment.
The modified Rankin Scale (mRS) | 30 days after onset
  Shift analysis of mRS scores at 30 days after onset. The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. (Score Description: 0---No symptoms at all. 1---No significant disability despite symptoms; able to carry out all usual duties and activities. 2---Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance. 3---Moderate disability; requiring some help, but able to walk without assistance. 4--- Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance. 5---Severe disability; bedridden, incontinent and requiring constant nursing care and attention. 6---Dead. The higher scores indicate worse functional disability and lower scores reflect better functional independence.
modified Rankin Scale (mRS) | 30 days after onset
  The rate of modified Rankin Scale (mRS) score > 3. The modified Rankin Scale (mRS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability. (Score Description: 0---No symptoms at all. 1---No significant disability despite symptoms; able to carry out all usual duties and activities. 2---Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance. 3---Moderate disability; requiring some help, but able to walk without assistance. 4--- Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance. 5---Severe disability; bedridden, incontinent and requiring constant nursing care and attention. 6---Dead. The higher scores indicate worse functional disability and lower scores reflect better functional independence.
Barthel Index (BI) score | 90-day follow-up visit
  Activities of daily living were evaluated using the Barthel Index (BI), a functional assessment scale ranging from 0 to 100, where higher scores indicate greater independence in daily activities and lower scores reflect more severe functional dependence.
All-cause mortality | 90-day follow-up visit
  Death caused by any reason.
Complication of severe dependent survival | 90-day follow-up visit
  eg, chest or other infections
Treated aneurysm rebleeding | 90-day follow-up visit
  Treated aneurysm rebleeding
Probable or definite bleed from another aneurysm | 90-day follow-up visit
  Probable or definite bleed from another aneurysm
Incidence of adverse events | 90-day follow-up visit
  Ischaemic stroke, Other intracranial haemorrhage, Cardiac, Cancer, Suicide, Renal failure, Infections not related to dependent survival, Other causes (eg, trauma, perforated ulcer, pulmonary embolus, neurodegenerative)

CONTACTS AND LOCATIONS:
Overall Officials: Renzhi Wang, MD, Study Chair — CUHK-Shenzhen; Xinyu Yang, Principal Investigator — CUHK-Shenzhen
Locations (1):
- School of Medicine Chinese University of Hong Kong-SHENZHEN, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Yang L, Yuan D, Luo Z, Li Y, Zhu X. The low-flow mask oxygen could be a more effective, comfortable, and easy-to-follow treatment for psychogenic hyperventilation syndrome: A double-blind, randomized controlled trial. Int Emerg Nurs. 2025 Aug;81:101636. doi: 10.1016/j.ienj.2025.101636. Epub 2025 Jun 17. PMID 40532319
- [Result] Darkwah Oppong M, Wrede KH, Muller D, Santos AN, Rauschenbach L, Dinger TF, Ahmadipour Y, Pierscianek D, Chihi M, Li Y, Deuschl C, Sure U, Jabbarli R. PaCO2-management in the neuro-critical care of patients with subarachnoid hemorrhage. Sci Rep. 2021 Sep 28;11(1):19191. doi: 10.1038/s41598-021-98462-2. PMID 34584136
- [Result] Cai G, Zhang X, Ou Q, Zhou Y, Huang L, Chen S, Zeng H, Jiang W, Wen M. Optimal Targets of the First 24-h Partial Pressure of Carbon Dioxide in Patients with Cerebral Injury: Data from the MIMIC-III and IV Database. Neurocrit Care. 2022 Apr;36(2):412-420. doi: 10.1007/s12028-021-01312-2. Epub 2021 Jul 30. PMID 34331211
- [Result] Su R, Li HL, Wang YM, Zhang L, Zhou JX. Association of dynamic changes in arterial partial pressure of carbon dioxide with neurological outcomes in aneurysmal subarachnoid hemorrhage. Heliyon. 2024 Oct 10;10(20):e39197. doi: 10.1016/j.heliyon.2024.e39197. eCollection 2024 Oct 30. PMID 39640813
- [Result] Carrera E, Schmidt JM, Fernandez L, Kurtz P, Merkow M, Stuart M, Lee K, Claassen J, Sander Connolly E, Mayer SA, Badjatia N. Spontaneous hyperventilation and brain tissue hypoxia in patients with severe brain injury. J Neurol Neurosurg Psychiatry. 2010 Jul;81(7):793-7. doi: 10.1136/jnnp.2009.174425. Epub 2009 Dec 3. PMID 19965840
- [Result] Coles JP, Fryer TD, Coleman MR, Smielewski P, Gupta AK, Minhas PS, Aigbirhio F, Chatfield DA, Williams GB, Boniface S, Carpenter TA, Clark JC, Pickard JD, Menon DK. Hyperventilation following head injury: effect on ischemic burden and cerebral oxidative metabolism. Crit Care Med. 2007 Feb;35(2):568-78. doi: 10.1097/01.CCM.0000254066.37187.88. PMID 17205016
- [Result] Coles JP, Minhas PS, Fryer TD, Smielewski P, Aigbirihio F, Donovan T, Downey SP, Williams G, Chatfield D, Matthews JC, Gupta AK, Carpenter TA, Clark JC, Pickard JD, Menon DK. Effect of hyperventilation on cerebral blood flow in traumatic head injury: clinical relevance and monitoring correlates. Crit Care Med. 2002 Sep;30(9):1950-9. doi: 10.1097/00003246-200209000-00002. PMID 12352026
- [Result] Robba C, Battaglini D, Abbas A, Sarrio E, Cinotti R, Asehnoune K, Taccone FS, Rocco PR, Schultz MJ, Citerio G, Stevens RD, Badenes R; ENIO collaborators. Clinical practice and effect of carbon dioxide on outcomes in mechanically ventilated acute brain-injured patients: a secondary analysis of the ENIO study. Intensive Care Med. 2024 Feb;50(2):234-246. doi: 10.1007/s00134-023-07305-3. Epub 2024 Jan 31. PMID 38294526
- [Result] Williamson CA, Sheehan KM, Tipirneni R, Roark CD, Pandey AS, Thompson BG, Rajajee V. The Association Between Spontaneous Hyperventilation, Delayed Cerebral Ischemia, and Poor Neurological Outcome in Patients with Subarachnoid Hemorrhage. Neurocrit Care. 2015 Dec;23(3):330-8. doi: 10.1007/s12028-015-0138-5. PMID 25846710